CLINICAL TRIAL: NCT06369402
Title: Cognitive Impairment and Cerebral Haemodynamics in Individuals With Symptomatic Peripheral Arterial Disease
Acronym: CInCH PAD
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0963
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-04

CONDITIONS: Peripheral Arterial Disease; Cognitive Impairment
MeSH Terms: conditions — Peripheral Arterial Disease; Cognitive Dysfunction | interventions — Ankle Brachial Index; Walk Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with symptomatic peripheral arterial disease: Individuals with intermittent claudication caused by confirmed peripheral arterial disease defined as a resting ankle-brachial pressure index of <0.9 and/or a post-exercise reduction in either ankle-brachial pressure index of >20% or absolute ankle pressure of >30mmHg.
  Interventions: Diagnostic Test: Cerebral haemodynamic testing using transcranial Doppler; Diagnostic Test: Ankle-brachial pressure index; Diagnostic Test: Six-minute walk test
- Healthy controls: Age- and sex-matched cohort of individuals without peripheral arterial disease.
  Interventions: Diagnostic Test: Cerebral haemodynamic testing using transcranial Doppler; Diagnostic Test: Ankle-brachial pressure index; Diagnostic Test: Six-minute walk test

INTERVENTIONS:
Diagnostic Test: Cerebral haemodynamic testing using transcranial Doppler — Measurement of cerebral haemodynamics using transcranial Doppler to insonate the middle cerebral arteries bilaterally testing neurovascular coupling with selected domains from the Addenbrooks cognitive examination III and the digit span forward and backwards.
Diagnostic Test: Ankle-brachial pressure index — Ratio of ankle to brachial blood pressure measured using handheld Doppler at rest and after exercise (six-minute walk test).
Diagnostic Test: Six-minute walk test — Supervised brisk walk for six minutes. Time and distance to onset of claudication pain and total distance walked (and total time walked if did not complete the full six minutes).

SUMMARY:
Background:

Arterial disease of the legs causes symptoms such as pain when walking and may ultimately lead to a leg amputation. Many older people with arterial disease of the legs also have problems with their thinking and memory. Blood flow in the brain may be altered in these people and may be a cause for memory and thinking problems.

Aim:

The aim of this project is to investigate whether people with arterial disease of the legs have altered blood flow in the brain causing problems with memory and thinking.

Research plan:

Twenty people with arterial disease of the legs causing pain while walking and twenty healthy people will have a series of non-invasive assessments. Arterial disease in the legs will be measured using ankle blood pressures before and after walking. Blood flow in the brain will be measured using ultrasound whilst performing memory and thinking tests. Results will be compared between the people with arterial disease in the legs and the healthy people to see if there are any differences in blood flow to the brain and memory and thinking.

Benefits to society:

This project will help determine if there is a link between arterial disease of the legs and memory and thinking problems caused by altered blood flow in the brain. It will enable future research in people with cognitive impairment caused by altered blood supply to the brain and to prevent confusion and further memory and thinking problems in people undergoing surgery for arterial disease of the legs.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide Informed volunteer/patient consent
* Male or female, aged ≥50 years of age
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* Good understanding of written and verbal English

Peripheral arterial disease specific inclusion criteria:

* Clinical diagnosis of symptomatic PAD (intermittent claudication) confirmed by positive haemodynamic tests (ABPI <0.90 in the symptomatic leg; and/or,
* Post-exercise [walk test] reduction in ABPI of >20% or post-exercise [walk test] reduction in absolute ankle pressure of >30mmHg)

Exclusion Criteria:

* Male or Female, aged under 50 years
* Pregnant
* Unable (in the Investigator's opinion) or unwilling to comply with any study requirements
* Major co-morbidity likely to affect cerebral autoregulation; severe respiratory disease, unilateral carotid artery stenosis (≥50%), atrial fibrillation, severe cardiac failure (left ventricular ejection fraction <20%), or extreme frailty
* History of significant diagnosed psychiatric disorder, learning disability (e.g. dyslexia) or neurological disorder (head injury, epilepsy, stroke and/or transient ischaemic attack [TIA])
* Diagnosis of dementia
* Uncorrected hearing impairment and/or significant visual impairment

Healthy control specific exclusion criteria

* Symptoms of intermittent claudication; and/or,
* Clinical diagnosis or history of PAD

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cohort of individuals with symptomatic peripheral arterial disease (intermittent claudication) with an age- and sex-matched healthy control cohort.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Peak % change of CBv from baseline | Baseline
  Change in response to performance of the ACE-III Cognitive Examination and Digit Span forward and backward.

SECONDARY OUTCOMES:
Autoregulation index (Tieck's model) | Baseline
  Change in response to performance of the ACE-III Cognitive Examination and Digit Span forward and backward.
Absolute score achieved on the Addenboook's cognitive examination (III) | Baseline
  Minimum score 0; Maximum score 100 (High scores indicate better cognitive performance)
Digit span forward and backward scores | Baseline
  Maximum list length correctly recalled and response consistency (total correct trials)

OTHER OUTCOMES:
Claudication distance | Baseline
  Distance to onset of pain in the six minute walk test
Maximal walking distance | Baseline
  Total distance walked during the six minute walk test
Ankle-brachial pressure index | Baseline
  Ratio of ankle blood pressure to the brachial blood pressure measured using handheld Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Rob D Sayers, MD, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Fully-anonymised electronic data will be stored in the Cerebral Haemodynamics in ageing and Stroke Medicine research database for 25 years and will be made available via the University of Leicester data repository (https://leicester.figshare.com/) for a minimum of 10 years.
Supporting Information: Study Protocol
Access Criteria: Access upon request to the study Chief Investigator (Prof R Sayers).
URL: https://leicester.figshare.com/